CLINICAL TRIAL: NCT01037621
Title: The Interaction of HSV-2 Co-infection in Veterans With Chronic Hepatitis C: the Effect of Valacyclovir on HCV Viral Load
Brief Title: Herpes Simplex Type 2 Co-infection in Veterans With Chronic Hepatitis C
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: G.V. (Sonny) Montgomery VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Wanda Hayes, Administrative Officer, Research and Development, G.V. (Sonny) Montgomery VA Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: VAL R 152; 2009-00348 (Other: G. V. Sonny Montgomery VAMC IRB)
Record Dates: First submitted 2009-12-22; First posted 2009-12-23 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Hepatitis C Virus Infection; Infection; Herpesvirus 2, Human
Keywords: Herpes simplex type 2; Hepatitis C virus; Valacyclovir; Herpes Simplex virus type 2 infection
MeSH Terms: conditions — Hepatitis C; Infections | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Valacyclovir — Valacyclovir 500 mg, 2 caplets twice daily for eight weeks
  Other Names: VALTREX

SUMMARY:
This trial is to determine the safety of valacyclovir in persons with chronic hepatitis C and herpes simplex type 2 infection. Participants will be randomized to valacyclovir or matching placebo. After receiving the initial therapy for eight weeks, the participants will cross over to the alternate therapy for an additional eight weeks. Each treatment period will be separated by a two-week period of daily placebo. The hypothesis is that treatment with valacyclovir will result in a significant reduction in serum levels of hepatitis C virus ribonucleic acid.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hepatitis C infection
* Clinical diagnosis of herpes simplex type 2 infection

Exclusion Criteria:

* HIV infection
* Other forms of chronic liver disease
* Chronic medical conditions
* On immunosuppressive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
The number of study participants who experience adverse events while receiving valacyclovir. | 18 weeks
  Tolerability assessments will be performed very two weeks while on study medications. Complete blood cell count, creatinine clearance and liver function tests will be performed every four weeks while on medications. Adverse events will be graded using the Division of AIDS Adverse Event Grading Table, Version 1.0, clarification August 2009. Based on previous clinical experience with valacyclovir, we expect the drug will be well-tolerated in patients with hepatitis C.

SECONDARY OUTCOMES:
The effect of valacyclovir compared with placebo to serum levels of HCV RNA | 18
  Serum HCV RNA will be measured at baseline and every four weeks while on study medication. We expect to see a decrease in HCV RNA >0.5 log10IU/mL during the valacyclovir phase compared with the placebo phase. The cross-over design will allow each patient to serve as their own control, providing data on the effect of HSV-2 suppression on HCV RNA.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jane Burton, M.D., Principal Investigator — G.V. (Sonny) Montgomery VA Medical Center
Locations (1):
- G.V. Sonny Montgomery VA Medical Center, Jackson, Mississippi, United States